CLINICAL TRIAL: NCT04015947
Title: Allogeneic Skin Grafting in the Treatment of Chronic Cutaneous Graft-versus-host Disease: a Pilot Study
Brief Title: Allogeneic Skin Grafting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DERM-2016-25255
Record Dates: First submitted 2018-08-07; First posted 2019-07-11 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: GVHD

STUDY DESIGN:
Intervention Model Description: This is an open label, single-institution pilot study to evaluate local response to split-thickness skin grafts from a matched bone marrow donor to chronic GVHD-affected skin in a hematopoietic stem cell transplant patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active treatment (Experimental): This is an open label, single-institution pilot study to evaluate local response to split-thickness skin grafts from a matched bone marrow donor to chronic GVHD-affected skin in a hematopoietic stem cell transplant patient.
  Interventions: Device: CelluTome® Epidermal Harvesting System

INTERVENTIONS:
Device: CelluTome® Epidermal Harvesting System — split-thickness skin grafts from a matched bone marrow donor using the CelluTome® Epidermal Harvesting System
  Other Names: split-thickness skin grafts

SUMMARY:
The primary study objective is to evaluate local response to split-thickness skin grafts from a matched bone marrow donor to chronic GVHD-affected skin in a hematopoietic stem cell transplant patient.

DETAILED DESCRIPTION:
While the mechanisms are still under active study, GVHD is thought to be a donor T-cell mediated attack that preferentially targets three organs: skin, intestine, and liver. T lymphocytes from the donor identify the patient's organ tissues as foreign and initiate inflammation, leading to end organ damage. The investigator's traditional approach has been to use immune suppressing drugs to dampen this inflammatory response after transplantation. However, this approach is ultimately ineffective for a significant percentage of patients. Therefore, the primary objective of this proposal is to test a novel non-immunosuppressive approach to treatment of cutaneous GVHD using allogeneic skin grafting in an effort to tolerize the engrafted immune system to skin it previously recognized as foreign. The potential benefit to transplant patients is tremendous, including reduced immunosuppression, improved quality of life and lower mortality.

A potential novel approach is to apply split-thickness skin grafts from the bone marrow donor to the affected patient's skin. There are four existing case reports that have shown positive outcomes in wound healing in chronic GVHD-associated ulcers. In all four cases, skin grafts were harvested from the patient's allogeneic HLA-matched sibling donors and placed over non-healing wounds (2-5). One case described global improvement in affected skin distant from the site of skin graft application, allowing for tapering of immunosuppressive medications. This suggests potential induction of tolerance by immune cells within the donated skin.

ELIGIBILITY:
Inclusion Criteria - Patient (Recipient)

* Subjects will be eligible to participate in the study if all of the following conditions exist:
* Diagnosis of chronic, sclerotic, cutaneous graft versus host disease with one or more areas of cutaneous sclerosis and
* More than 1 year after HCT with stable hematopoietic engraftment and original transplant donor is available and agrees to be the epidermal donor for this study
* Stable (mixed or full) donor hematopoietic engraftment
* Original transplant donor is available and willing to be the epidermis donor
* Site for skin grafting free of cellulitis or other evidence of infection
* Insurance pre-authorization for procedure
* Voluntary written consent prior to any research related procedures or treatment.

Inclusion Criteria - Donor

* Age > 18 years (based on prior safety testing of the device)
* Healthy on physical examination in the opinion of the evaluating physician
* Known negativity for Hepatitis B and C, HIV, and HTLV1/2
* Voluntary written consent prior to any research related procedures

Exclusion Criteria

Subjects will be excluded from participation in the study if any of the following conditions exist:

* Patient with cutaneous infection
* Patient with recent change in medical management of chronic cutaneous GVHD (new medication or therapy, or change in dosing of existing medication) within one month of start date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in CGAA | Change from baseline up to 12 months
  Evaluation of clinical improvement in inflammation and sclerosis based on visual inspection and photodocumentation with outcome outcomes determined using the Chronic GVHD Activity Assessment (CGAA) to measure therapeutic response. The CGAA is an 8-item assessment measuring symptom severity of GVHD on a scale from 0 (not present) to 10 (as bad as you can imagine). Global score is calculated by summing items.
Change in ELISA Markers of GVHD | Change from baseline up to 12 months
  Chronic GVHD lesions will be assessed following transplantation through serum ELISA assays of elafin and CXCL10 (validated biomarkers for assessment of GVHD disease activity)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No